CLINICAL TRIAL: NCT02691260
Title: Incentivizing Behavior Change Skills to Promote Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00056410; 1R34HL125669-01A1 (NIH)
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Obesity
Keywords: obesity; behavioral intervention; diet
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- no incentives (No Intervention): Participants do not receive financial incentives.
- incentives for dietary self-monitoring (Active Comparator): Participants receive financial incentives for dietary self-monitoring.
  Interventions: Behavioral: incentives for dietary self-monitoring
- incentives for interim weight loss (Active Comparator): Participants receive financial incentives for interim weight loss.
  Interventions: Behavioral: incentives for interim weight loss
- incentives for both (Experimental): Participants receive incentives for dietary self-monitoring and interim weight loss.
  Interventions: Behavioral: incentives for both

INTERVENTIONS:
Behavioral: incentives for dietary self-monitoring — Participants will receive intermittent financial incentives for recording their dietary intake on a dietary mobile phone application.
  Arms: incentives for dietary self-monitoring
Behavioral: incentives for interim weight loss — Participants will receive intermittent financial incentives for losing an expected amount of weight based weight obtained weekly.
  Arms: incentives for interim weight loss
Behavioral: incentives for both — Participants will receive intermittent financial incentives for recording their dietary intake on a dietary mobile phone application and for losing an expected amount of weight based on weight obtained weekly.
  Arms: incentives for both

SUMMARY:
The purpose of this study is to determine the feasibility of providing incentives to people enrolled in a weight-loss program for dietary self-monitoring and/or interim weight loss.

DETAILED DESCRIPTION:
In this study, community outpatients will participate in an effective, 24-week, low-carbohydrate weight loss program delivered via biweekly group classes. An innovative information technology (IT) solution will collate dietary self-monitoring data (input by patients via a mobile phone dietary application) and weight loss data (input by patients via remote scale). An algorithm will classify participants as achieving adequate or inadequate dietary self-monitoring and weight loss to earn intermittent rewards of varying value in real-time. Participants will be notified of earning rewards via text messaging.

ELIGIBILITY:
Inclusion Criteria:

* desire to lose weight;
* agree to attend visits per protocol;
* access to telephone and transportation;
* English speaking;
* able to complete study measures;
* smart phone with data and texting plan;
* body mass index 30 kg/m2 or greater

Exclusion Criteria:

* pregnancy, breastfeeding, or lack of birth control if premenopausal
* dementia, excessive alcohol use, or psychiatric illness
* weight loss >4.5 kg in month prior to screening
* weight > 380 lb (due to limit of cellular scale)
* enrollment in other weight loss program
* residing in nursing home or receiving home health care
* unable to attend weight loss group at scheduled times
* impaired hearing
* medication other than metformin, incretin mimetics and incretin enhances for type 2 diabetes
* unstable heart disease in 3 months prior to screening
* furosemide 40 mg or higher (or equivalent)
* chronic kidney disease
* 2 or more errors on cognitive screener
* blood pressure ≥160/100 mmHg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-04; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Shaw, PhD, RN, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Voils CI, Levine E, Gierisch JM, Pendergast J, Hale SL, McVay MA, Reed SD, Yancy WS Jr, Bennett G, Strawbridge EM, White AC, Shaw RJ. Study protocol for Log2Lose: A feasibility randomized controlled trial to evaluate financial incentives for dietary self-monitoring and interim weight loss in adults with obesity. Contemp Clin Trials. 2018 Feb;65:116-122. doi: 10.1016/j.cct.2017.12.007. Epub 2017 Dec 28. PMID 29289702
- [Derived] Gavin KL, Almeida EJ, Voils CI, Crane MM, Shaw R, Yancy WS Jr, Pendergast J, Olsen MK. Comparison of weight captured via electronic health record and cellular scales to the gold-standard clinical method. Obes Sci Pract. 2023 Jan 12;9(4):337-345. doi: 10.1002/osp4.656. eCollection 2023 Aug. PMID 37546286
- [Derived] Voils CI, Pendergast J, Hale SL, Gierisch JM, Strawbridge EM, Levine E, McVay MA, Reed SD, Yancy WS, Shaw RJ. A randomized feasibility pilot trial of a financial incentives intervention for dietary self-monitoring and weight loss in adults with obesity. Transl Behav Med. 2021 Apr 26;11(4):954-969. doi: 10.1093/tbm/ibaa102. PMID 33245118
- [Derived] Shaw R, Levine E, Streicher M, Strawbridge E, Gierisch J, Pendergast J, Hale S, Reed S, McVay M, Simmons D, Yancy W, Bennett G, Voils C. Log2Lose: Development and Lessons Learned From a Mobile Technology Weight Loss Intervention. JMIR Mhealth Uhealth. 2019 Feb 13;7(2):e11972. doi: 10.2196/11972. PMID 30758297

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | no Incentives | Incentives for Dietary Self-monitoring | Incentives for Interim Weight Loss | Incentives for Both
Started | 26 | 26 | 27 | 26
Completed | 24 | 24 | 25 | 23
Not Completed | 2 | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | no Incentives | Incentives for Dietary Self-monitoring | Incentives for Interim Weight Loss | Incentives for Both | Total
Number analyzed (Participants) | 26 | 26 | 27 | 26 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 26 | 24 | 92
  >=65 years | 4 | 6 | 1 | 2 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.65 (12.73) | 51.27 (15.46) | 46.44 (11.15) | 45.92 (12.84) | 48.3 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 21 | 25 | 92
  Male | 4 | 2 | 6 | 1 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 26 | 26 | 27 | 23 | 102
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 12 | 8 | 33
  White | 15 | 19 | 13 | 17 | 64
  More than one race | 3 | 0 | 2 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 26 | 27 | 26 | 105

OUTCOME MEASURES:

1. Primary Outcome: Weight Change From Baseline to 24 Weeks
Description: Measured in pounds
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Pounds (lbs.)
Arm/Group | no Incentives | Incentives for Dietary Self-monitoring | Incentives for Interim Weight Loss | Incentives for Both
Number analyzed (Participants) | 24 | 24 | 25 | 23
Pounds (lbs.) | -8.046 (13.316) | -15.496 (15.391) | -12.167 (17.884) | -17.696 (10.312)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were also collected during in-person visits
Arm/Group | no Incentives | Incentives for Dietary Self-monitoring | Incentives for Interim Weight Loss | Incentives for Both
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/26 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 3/26 | 3/26 | 5/27 | 1/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | no Incentives (N=26) | Incentives for Dietary Self-monitoring (N=26) | Incentives for Interim Weight Loss (N=27) | Incentives for Both (N=26)
Hospitalization (Gastrointestinal disorders) | 1 (26) | 0 (0) | 0 (0) | 0 (0) — Infected gallbladder removed. Preceding study: Diagnosed with IBS for 20 yrs, GERD longstanding, upper abdomen pains intermittently for >1year. Possible high fat diet was related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | no Incentives (N=26) | Incentives for Dietary Self-monitoring (N=26) | Incentives for Interim Weight Loss (N=27) | Incentives for Both (N=26)
Swollen lymph node (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dog bite (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Generally unwell (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Felt weak, flushed and 'generally unwell'. Participant then decided to add carbs back into diet and stated that she felt better once she incorporated carbs back into her diet.
Gout like symptoms (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ER visit for allergies (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ate peanuts while traveling and irritated diverticulitis
irritated diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ate popcorn as snack, it irritated diverticulitis
Planned foot surgery (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Weight adjustment 4 to 6 pound increase with cast consideration
Bone achiness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
High blood pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
blood in urine (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pt stopped diet upon recommendation from physician
erythema (Immune system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) — erythema on facial areas. Participant experienced this before but flared up since beginning diet.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT02691260/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT02691260/Prot_SAP_001.pdf